

# Assessing Breast Cancer Risk Prior to Gender-Affirming Chest Masculinization Surgery in Transgender Men

Short Title

BC Risk Assessment Before Top Surgery

Study Principal Investigator Chandler Cortina, MD, MS

Version 1.0 01/30/2023

#### **Proprietary and Confidential**

The information in this document is considered privileged and confidential and may not be disclosed to others except to the extent necessary to obtain Institutional Review Board approval and informed consent, or as required by federal and state laws. Persons to whom this information is disclosed should be informed that this information is privileged and confidential and that it should not be further disclosed.

#### STUDY AND CONTACT INFORMATION

Protocol Long Title: Assessing Breast Cancer Risk Prior to Gender-Affirming Chest

Masculinization Surgery in Transgender Men

MCW Protocol No.: PRO00045830

#### **Principal Investigator:**

Chandler Cortina, MD, MS Assistant Professor of Surgery Division of Surgical Oncology Medical College of Wisconsin 9200 W. Wisconsin Ave. Milwaukee, WI 53226 Phone: 414-805-1400

Email: ccortina@mcw.edu

#### Co-investigator:

Kristen Klement, MD Assistant Professor of Plastic Surgery Medical College of Wisconsin 1155 N. Mayfair Rd.

Milwaukee, WI 53226 Phone: 414-955-1000 Email: kklement@mcw.edu

## Co-investigator:

Sarah Sasor, MD

Assistant Professor of Plastic Surgery

Medical College of Wisconsin

1155 N. Mayfair Rd. Milwaukee, WI 53226 Phone: 414-955-1000 Email: ssasor@mcw.edu

#### Statistician:

Ruta Brazauskas, PhD Associate Professor of Biostatistics Institute for Health and Equity Medical College of Wisconsin 8701 Watertown Plank Rd. Milwaukee, WI 53226

Phone: 414-955-8687 Email: ruta@mcw.edu

#### **Funding Source:**

Advancing a Healthier Wisconsin Endowment

#### Co-investigator:

Erin Doren, MD, MPH Associate Professor of Plastic Surgery

Medical College of Wisconsin

1155 N. Mayfair Rd. Milwaukee, WI 53226 Phone: 414-955-1000 Email: edoren@mcw.edu

#### Co-investigator:

Kate Krucoff, MD

Assistant Professor of Plastic Surgery

Medical College of Wisconsin 9200 W. Wisconsin Ave. Milwaukee, WI 53226 Phone: 414-955-3860 Email: kkrucoff@mcw.edu

#### Co-investigator

Anna Purdy, APNP

Nurse Practitioner, Department of Surgery

Division of Surgical Oncology Medical College of Wisconsin 9200 W. Wisconsin Ave. Milwaukee, WI 53226

Phone: 414-955-1428 Email: <a href="mailto:apurdy@mcw.edu">apurdy@mcw.edu</a>

#### **Medical Geneticist (Collaborator):**

Samantha Stachowiak, MS, CGS Certified Genetic Counselor Medical College of Wisconsin 9200 W Wisconsin Ave Milwaukee, WI 53226 Phone: 414-955-4222

Email: sstachowiak@mcw.edu

Version No.: 1.0

# **TABLE OF CONTENTS**

| STUDY | AND CONTACT INFORMATION | 2 |
|---|---|---|
| TABLE | OF CONTENTS | 3 |
| PROTO | COL SUMMARY | 5 |
| STUDY | SCHEMA | 7 |
| STUDY | CALENDAR | 8 |
| LIST OF | ABBREVIATIONS | 9 |
| 1.0 | BACKGROUND | 10 |
| 1.1 | Breast Cancer in Transgender and Nonbinary Persons | 10 |
| 1.2 | Rationale | 11 |
| 2.0 | OBJECTIVES AND ENDPOINTS | 12 |
| 2.1 | Primary Objectives | 12 |
| 2.2 | Primary Endpoints | 12 |
| 3.0 | SUBJECT POPULATION AND ELIGIBILITY | 12 |
| 3.1 | Subject Population | 12 |
| 3.2 | Eligibility Criteria | 12 |
| 4.0 | ACCRUAL GOAL AND STUDY DURATION | 13 |
| 5.0 | PATIENT RECRUITMENT AND REGISTRATION | 13 |
| 6.0 | STUDY DESIGN, PROCEDURES, AND MEASUREMENTS | |
| 6.1 | Overview of the Study Design Workflow | 14 |
| 6.2 | Visit 1: Breast Cancer Risk Assessment, Risk Categorization, and Initial Counseling | , 14 |
| 6.3 | Breast Cancer Genetic Testing | 15 |
| 6.4 | Visit 2: Surgical Risk-Reducing Mastectomy Counseling | 16 |
| 6.5 | Data Factors | 16 |
| 7.0 | SUBJECT WITHDRAWAL, END OF STUDY, AND STUDY DISCONTINUATION | 17 |
| 7.1 | Subject Withdrawal | 17 |
| 7.2 | End of Study Definition | 18 |
| 7.3 | Study Discontinuation and Closure | 18 |
| 8.0 | ADVERSE EVENTS: DEFINITIONS, COLLECTION, AND REPORTING | 18 |
| 8.1 | Definitions | 18 |
| 8.2 | Collection and Reporting Requirements for Adverse Events and Serious Adverse Events | 20 |
| 8.3 | Unanticipated Problem Involving Risk to Subject or Other (UPIRSO) | 20 |
| 8.4 | Subject Complaints | 20 |


| 9.0 | STATISTICAL CONSIDERATIONS | 21 |
|---|---|---|
| 9.1 | Sample Size Determination and Accrual Estimates | 21 |
| 9.2 | Analysis Plan | 21 |
| 9.3 | Missing Data | 21 |
| 10.0 | DATA AND SAFETY MONITORING PLAN (DSMP) | 21 |
| 10.1 | Data and Safety Management Overview | 21 |
| 10.2 | Study Team | 22 |
| 10.3 | Quality Assurance | 22 |
| 10.4 | DSMC | 22 |
| 11.0 | REGULATORY COMPLIANCE, ETHICS, AND STUDY MANAGEMENT | 23 |
| 11.1 | Ethical Standard | 23 |
| 11.2 | Regulatory Compliance | 23 |
| 11.3 | Informed Consent Process | 23 |
| 11.4 | Subject Confidentiality and Access to Source Documents/Data | 23 |
| 11.5 | Risk-Benefit Assessment | 24 |
| 11.6 | Protection of Human Subjects | 24 |
| 11.7 | Changes in the Protocol | 25 |
| 11.8 | Investigator Compliance | 25 |
| 12.0 | DATA MANAGEMENT | 26 |
| 12.1 | Data Management Plan | 26 |
| 12.2 | Disseminating and Publishing Data | 26 |
| REFERE | ENCES | 27 |
| APPENI | DIX 1. Lifetime Breast Cancer Risk Assessment Form | 32 |
| | DIX 2. NCCN Testing Criteria for High-Penetrance Breast And/Or Ovarian Cancer ibility Genes | 33 |


# **PROTOCOL SUMMARY**

| Title | Assessing Breast Cancer Risk Prior to Gender-Affirming Chest Masculinization Surgery in Transgender Men |
|---|---|
| Principal Investigator | Chandler Cortina, MD, MS |
| Study Sites | Froedtert Health and the Medical College of Wisconsin |
| Study Population | Non-cisgender adults seeking chest masculinization surgery (top surgery). |
| Primary Objectives | <ol> <li>To determine the prevalence of TGNB persons undergoing chest masculinization surgery who have an elevated lifetime risk of breast cancer development and prevalence of those who undergo genetic counseling.</li> <li>To determine whether those TGNB persons at elevated risk of breast cancer development choose to undergo risk-reducing mastectomies as part of their chest masculinization surgery.</li> <li>To assess and compare the self-perceived breast cancer risk with calculated risk.</li> </ol> |
| Primary Endpoints | <ol> <li>The percentage of all participants undergoing chest masculinization surgery who are at elevated lifetime risk of BC development (<i>i.e.</i>, &gt;17%) and those who undergo genetic counseling. Lifetime BC risk will be estimated utilizing the Gail and IBIS models.</li> <li>The percentage of those participants with moderate to high lifetime BC risk or pathogenic germline variant that say they would choose to undergo a risk-reducing mastectomy.</li> <li>The accuracy of self-perceived BC risk, as measured by the Visual Analog Scale (VAS), and the personalized BC risk assessment taken after the VAS.</li> </ol> |
| Main Eligibility Criteria | <ul> <li>≥18 years old.</li> <li>Assigned female or intersex at birth and identify as non-cisgender.</li> <li>Considering undergoing gender-affirming chest masculinization surgery.</li> <li>Ability to communicate in English.</li> <li>Ability to understand a written informed consent document, and the willingness to sign it.</li> </ul> |
| Study Design | Prospective, single-arm interventional pilot study designed to test whether a breast cancer risk assessment, genetic testing (when applicable), and surgical oncologist consultation can inform those TGNB patients at elevated risk for breast cancer development to undergo risk-reducing mastectomies in tandem with their gender-affirming chest masculinization surgery. |


| Intervention | Breast cancer risk assessment and education. |
|---|---|
| Number of Subjects | 35 patients (100 patients screened) |
| Subject Participation<br>Duration | Breast cancer risk assessment will take approximately 30 minutes. Additionally, we wish to follow participants via record review for up to 1 year. |
| Estimated Time to Complete Enrollment | One year |


#### STUDY SCHEMA




#### STUDY CALENDAR

| Assessments and Procedures | Screening/<br>Enrollment | Visit 1 | Cancer<br>Genetics<br>Clinic<br>Visit <sup>b</sup> | Visit 2 <sup>c</sup> | Follow-up <sup>d</sup> |
|---|---|---|---|---|---|
| | Day -60 to -1 | Day +1 | | | |
| Eligibility Confirmation | X | | | | |
| Informed Consent | Х | Xa | | | |
| Patient Registration | Х | Xa | | | |
| Visual Analog Scale | | Х | | | |
| Personalized BC Risk<br>Assessment (Gail and/or<br>IBIS model) | | Х | | | |
| Genetic Counseling <sup>b</sup> | | | Xp | | |
| Genetic Testing <sup>b</sup> | | | Xp | | |
| Surgical Oncologist Risk-<br>Reducing Mastectomy<br>Counseling Session <sup>o</sup> | | | | Xc | |
| Data Collection | | Х | Х | Х | Х |
| Adverse Events Collection | | Х | Х | Х | |

#### **Footnotes**

- <sup>a</sup> During Visit 1, the study team will be available to answer any additional questions the potential participant may have about the study and confirm whether they were consented. If not done so already and as an option, a potential participant will have the opportunity to sign the informed consent form in person.
- b Only those study participants with a family history suggestive of a pathogenic variant and/or with an elevated breast cancer risk who meet genetic testing guidelines (Appendix 2)<sup>1, 2</sup> will be referred to the Cancer Genetics Clinic to undergo a formal genetic counseling session and possible germline genetic testing. Genetic testing will be performed via the Ambry Genetics® Panel per institutional standards. See Section 6.3 for additional details.
- Only those study participants with an estimated lifetime breast cancer risk >17% (defined by the Gail model [https://ibis.ikonopedia.com] and/or IBIS model [https://www.mdcalc.com/calc/3647/gail-model-breast-cancer-risk]) or with a pathogenic germline mutation known to increase breast cancer risk will be offered to meet with the PI to discuss the utility of considering risk-reducing mastectomies as part of their chest masculinization surgery. If a subject is referred to the Cancer Genetics Clinic, Visit 2 is to occur after their Cancer Genetics Clinic visit.
- <sup>d</sup> Participants with an estimated lifetime breast cancer risk >17% may be followed-up once within 60 days after the end of the funding period to determine if they either (i) underwent their chest masculinization surgery with or without the risk-reducing mastectomies, (ii) scheduled but did not undergo their chest masculinization surgery with or without the risk-reducing mastectomies, or (iii) say they would choose to schedule/undergo risk-reducing mastectomies as part of their chest masculinization surgery. Regarding (i) and (ii), follow-up data will only be collected from participants that had their procedure(s) performed by a MCW Plastic Surgery team member (study Co-Is) and, in certain instances, the study PI.


#### LIST OF ABBREVIATIONS

AE adverse event
BC breast cancer
CDH1 cadherin 1

CFR Code of Federal Regulations

CHEK2 checkpoint kinase 2
Co-I Co-investigator

CTCAE Common Terminology Criteria for Adverse Events

CTEP Cancer Therapy Evaluation Program

CTO Clinical Trials Office

CTSI Clinical and Translational Science Institute
DSMC Data and Safety Monitoring Committee

DSMP Data and Safety Monitoring Plan

FH Froedtert Health System
GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act
IBIS Tyrer-Cuzick Breast Cancer Risk Evaluation Tool

ICH International Council for Harmonisation

ICMJE International Committee of Medical Journal Editors

IRB Institutional Review Board MCW Medical College of Wisconsin

MCWCC Medical College of Wisconsin Cancer Center

MRI magnetic resonance imaging
NCI National Cancer Institute

PALB2 partner and localizer of BRCA2
PHI protected health information

PI Principal Investigator

PTEN phosphatase and tensin homolog

SAE serious adverse events

SOP standard operating procedure SRC Scientific Review Committee

TGNB transgender and nonbinary persons

US United States

#### 1.0 BACKGROUND

#### 1.1 Breast Cancer in Transgender and Nonbinary Persons

The population of transgender and nonbinary persons (TGNB) in Wisconsin and the United States (US) is steadily increasing and as this population grows, the number of individuals seeking gender-affirming therapies, including gender-affirming operations and gender-affirming hormone therapy, is also increasing.<sup>3-5</sup> In calendar year 2021 alone, the Froedtert & Medical College of Wisconsin Inclusion Health Clinic cared for >700 TGNB persons, and this patient population has been steadily increasing since the clinic opened in 2018. An example of gender-affirming surgery is chest masculinization surgery, colloquially called top surgery, in which the majority of breast tissue is removed in a person with a female sex assigned at birth to allow the chest to appear masculine.<sup>6</sup> While chest masculinization surgery removes most glandular breast tissue, some

breast tissue is often left behind to allow for appropriate cosmetic contouring of the chest (Figure 1) and is not considered synonymous to an risk-reducing oncologic mastectomy.6, 7 An oncologic risk-reducing mastectomy seeks to remove all breast tissue in an effort to minimize the future risk of breast cancer



Figure 1. Before (A) and after (B) photos of a TGM after chest masculinization surgery

(BC) development in persons with an elevated lifetime risk of breast cancer.<sup>8-10</sup> Additionally, there is an increasing number of reported cases of TG men developing BC after chest masculinization surgery, secondary to the lack of data to support routine personalized BC risk assessment prior to chest masculinization surgery or for BC screening after chest masculinization surgery.<sup>7, 11-14</sup> Although gender-affirming therapies are associated with improved mental health outcomes and well-being for TGNB persons,<sup>15</sup> the potential long-term effects of these therapies on overall health, including future breast cancer risk, are not well understood.<sup>16-18</sup>

BC is the most common non-skin cancer in cisgender women. The current average lifetime risk for cisgender women is approximately 13% for a person who lives to be age 85 years in the United States. 19, 20 A person's lifetime risk of BC development may be dramatically impacted by a family history of BC, increased breast density, a personal history of atypical hyperplasia, lobular carcinoma in situ, high-dose radiation to the chest before age 30, or inherited genetic mutations in BC susceptibility genes.<sup>21-29</sup> Two well-validated models have been developed to estimate an individual's personalized percent lifetime BC risk: the Gail Model<sup>30-36</sup> and the Tyrer-Cuzick BC Risk Evaluation Tool (also called IBIS) that incorporate personal history (e.g., first age at menarche, history of breast biopsies) and family breast and ovarian cancer history to calculate future breast cancer risk compared to the average cisgender woman. 37-43 Both models provide a percent estimate of a person's lifetime risk compared to the average women (ex: 35% lifetime risk for a person compared to 12.5% for average risk peer). Cisqender women with a moderate lifetime BC risk (17%-30%)<sup>44</sup> can be offered BC screening at an younger age (prior to age 40 years), enhanced BC screening with magnetic resonance imaging (MRI), or risk-reducing medications such as tamoxifen or raloxifene. 45-49 Those with a high lifetime BC risk, defined as >30%, 44 can be offered the previous options and may also consider risk-reducing mastectomies, a procedure reserved for this group given its potential risks and complications. 1, 9, 50-52 High and moderate penetrant pathogenic variants (BRCA1/2, PTEN, CDH1, PALB2, CHEK2, ATM, etc.) are known to elevate BC risk.<sup>2, 53-57</sup> Pathogenic variants (mutations) may be found through exploratory

processes, such as commercially available kits like 23andMe<sup>®</sup>, or through formal evaluation by a healthcare provider based on personal or family history. Risk-reducing mastectomies are generally offered to persons with a known pathogenic variant or a lifetime BC risk >30%.<sup>8, 58, 59</sup> While the ability to reduce BC incidence in these populations with risk-reducing mastectomies is well documented, there is insufficient data to determine if the operation provides a clear mortality benefit, with the exception of persons with a BRCA1 mutation.<sup>8, 9, 50, 58, 59</sup>

Self-perceived BC risk has the potential to influence risk-modifying behaviors such as alcohol and smoking use, uptake of cancer screening recommendations, and has been demonstrated to influence the decision for risk-reducing mastectomies in cisgender women with an elevated lifetime BC risk. 60-62 There is no contemporary data on perceived BC risk prior to chest masculinization surgery in TGNB persons, which may potentially influence an individual's decision to undergo chest masculinization surgery ± risk-reducing mastectomies. Given that an increasing number of TGNB persons are undergoing gender-affirming chest masculinization surgery and that no data exists on the operation's ability to reduce the incidence of BC, a clear opportunity exists to perform routine personalized BC risk assessment (± genetic testing) prior to chest masculinization surgery to identify those persons with a high lifetime BC risk who may benefit from undergoing oncologic risk-reducing mastectomies as part of their gender-affirming chest masculinization surgery. 63 Currently, these individuals do not undergo personalized BC risk assessment prior to chest masculinization surgery. Additionally, there is a need to examine both the accuracy of self-perceived BC risk in TGNB persons and how it may influence genderaffirming surgical decision making. Understanding BC risk in TGNB persons is a critical step in mitigating cancer disparities in this underserved population in Wisconsin and across the United States and to ensure patients are informed of this risk prior to undergoing chest masculinization surgery.

The Froedtert & MCW Inclusion Health Clinic opened in July 2018 and is located on the Milwaukee Regional Medical Center grounds within the Sargeant Health Center. The clinic is focused on providing health care for LGBTQ+ individuals. Services include primary and preventive care, obstetrics and gynecology, HIV prevention, gender-affirming care, and psychiatric care. The clinics are the only ones of its kind in Wisconsin and in the 2020-2021 fiscal year, cared for >1,600 individual patients, of which >600 identify as transgender. The unique relation with the Inclusion Health Clinic, the Southeastern Wisconsin LGBTQ+ community, and a skilled Plastic Surgery team allow for a unique opportunity to conduct this investigation.

#### 1.2 Rationale

The goals of this pilot study are to 1) determine the percent of TGNB persons undergoing chest masculinization surgery who have an elevated lifetime risk of BC development (>17%) or a pathogenic genetic mutation that increased the risk of BC development (BRCA1/2, ATM, etc.), 2) measure the percent who are at risk and say they would choose to undergo risk-reducing mastectomies as part of chest masculinization surgery, and 3) assess and compare self-perceived BC risk with calculated risk. The results of this study will substantially inform TGNB patients and surgeons on the utility of personalized BC risk assessment prior to chest masculinization surgery and the accuracy of self-perceived BC risk in TGNB persons. This project has the potential to set a new standard of care that all TGNB persons should undergo a personalized BC risk assessment prior to gender-affirming surgery.


#### 2.0 OBJECTIVES AND ENDPOINTS

This prospective, single-arm interventional pilot study is designed to test whether a breast cancer risk assessment, genetic testing (when applicable), and surgical oncologist consultation can inform those TGNB patients at elevated risk for breast cancer (BC) development to undergo risk-reducing mastectomies in tandem with their gender-affirming chest masculinization surgery. This study is expected to collect and analyze novel data that describes the prevalence of elevated BC risk in the TGNB population and the concordance between self-perceived BC risk and calculated risk, a pressing need for which little is known.

#### 2.1 Primary Objectives

- 1. To determine the prevalence of TGNB persons undergoing chest masculinization surgery who have an elevated lifetime risk of breast cancer development and prevalence of those who undergo genetic counseling.
- 2. To determine whether those TGNB persons at elevated risk of breast cancer development choose to undergo risk-reducing mastectomies as part of their chest masculinization surgery.
- 3. To assess and compare the self-perceived breast cancer risk with calculated risk.

#### 2.2 Primary Endpoints

- 1. The percentage of all participants undergoing chest masculinization surgery who are at elevated lifetime risk of BC development (*i.e.*, >17%) and those who undergo genetic counseling. Lifetime BC risk will be estimated utilizing the Gail and IBIS models.
- The percentage of those participants with moderate to high lifetime BC risk or pathogenic germline variant that say they would choose to undergo a risk-reducing mastectomy.
- 3. The accuracy of self-perceived BC risk, as measured by the Visual Analog Scale (VAS), and the personalized BC risk assessment taken after the VAS.

#### 3.0 SUBJECT POPULATION AND ELIGIBILITY

MCW must follow all MCW IRB requirements and policies regarding subject participation, found here: <a href="https://www.mcw.edu/HRPP/Policies-Procedures.htm">https://www.mcw.edu/HRPP/Policies-Procedures.htm</a>

#### 3.1 Subject Population

Non-cisgender adults seeking chest masculinization surgery (top surgery).

#### 3.2 Eligibility Criteria

The study team will evaluate eligibility according to the following criteria. Subjects must meet <u>all</u> inclusion and <u>none</u> of the exclusion criteria to be registered on to the study. Any questions or concerns regarding eligibility should be directed to the PI, Dr. Chandler Cortina (ccortina@mcw.edu).

No waivers of protocol eligibility will be granted.

#### 3.2.1 Inclusion Criteria

A potential study subject who meets <u>all</u> of the following inclusion criteria is <u>eligible</u> to participate in the study.

- 1. ≥18 years old.
- 2. Assigned female or intersex at birth and identify as non-cisgender.
- 3. Any individual considering undergoing gender-affirming chest masculinization surgery
- 4. Ability to communicate in English.
- 5. Ability to understand a written informed consent document, and the willingness to sign it.

#### 3.2.2 Exclusion Criteria

A potential study subject who meets <u>any</u> of the following exclusion criteria is <u>ineligible</u> to participate in the study.

- 1. <18 years old.
- 2. Assigned male sex at birth.
- 3. Previously underwent chest masculinization surgery or any form of oncological mastectomy for the purposes of risk-reduction or cancer treatment.
- 4. Any previous or current history of breast cancer, including ductal carcina in situ (DCIS).
- 5. Inability to communicate in English.

#### 4.0 ACCRUAL GOAL AND STUDY DURATION

The Froedtert and MCW Plastic Surgery Clinics see 75-100 individuals seeking top surgery per year. In 2022, MCW Plastic Surgeons performed 55 chest masculinization operations. Based on our study protocol and budget allotment, we expect to screen 100 patients and recruit 35 participants for this study.

The study is estimated to reach completion approximately 12 months from the time the study opens to accrual.

#### 5.0 PATIENT RECRUITMENT AND REGISTRATION

TGNB individuals seen in the Plastic Surgery Clinic for surgical consultation for gender-affirming chest masculinization surgery will be given the opportunity to participate in the study. The PI or Anna Purdy, APNP will review the Plastic Surgeons' schedules to notify plastic surgeons of potential eligible participants. Patients will be provided a flyer that provides an overview of the study premise, measures, and study team contact information.


Once an individual confirms interest in the study, they will be screened by the PI for eligibility through Epic and then contacted via phone and/or email to discuss the study, answer any question, and the potential participant will be provided with an electronic and encrypted copy of the study's consent form, if interested in participating. Participants may provide their electronic signature and emailed back to the PI prior to Visit 1, at the time of Visit 1, or if meeting in person can provide a written signature.

Eligible participants who want to participate will be scheduled for a 30-minute appointment (Visit 1) in the Breast Care Clinic, located within the Froedtert and Medical College of Wisconsin Clinical Cancer Center, with either Anna Purdy, APNP or the PI. Eligible participants will also be given the given the option to have only a telephone or virtual visit (at the individuals' discretion). Patients who wish to meet in person for this screening assessment will be billed for services if seen formally in-person in the Breast Care Clinic. Participants will be incentivized to participate by receiving a \$100 gift card.

## 6.0 STUDY DESIGN, PROCEDURES, AND MEASUREMENTS

#### 6.1 Overview of the Study Design Workflow



<sup>\*</sup>Activities that occur after the personalized BC risk assessment are participant choice, standard practice, and will be collected as part of study data.

# 6.2 Visit 1: Breast Cancer Risk Assessment, Risk Categorization, and Initial Counseling

Participants will be scheduled within 60 days of initial screening and consent to undergo a personalized BC risk assessment utilizing the Gail and IBIS tools, which are both validated and widely used assessments. 37-43 During Visit 1, participants will identify their self-perceived lifetime BC risk on the Visual Analog Scale (Appendix 1) as part of the initial study intake, which will also acquire identifiable patient data (name, date of birth, and medical record number) and demographic information (race, ethnicity, age, sex assigned at birth, gender, etc; see Section 6.5 for a comprehensive list of data factors to be collected). The PI and Anna Purdy, APNP will enter the risk estimates from the Gail (https://ibis.ikonopedia.com) **IBIS** and

(<u>https://www.mdcalc.com/calc/3647/gail-model-breast-cancer-risk</u>) models into the same intake form, and calculate the mean BC calculated risk as the average of the two models:

$$\textit{Mean Lifetime BC Risk} = \frac{\textit{Risk from Gail Model} + \textit{Risk from IBIS Model}}{2}$$

For participants <35 years old, in which Gail is not validated, only the IBIS lifetime BC risk will be used, and a mean lifetime risk will *not* be calculated.

Participants with an **average** lifetime BC risk, defined as ≤17%,<sup>44</sup> will be recommended to continue their gender-affirming operation as planned and will not be scheduled for a second visit.

Those with a **moderate** lifetime BC risk, defined as 17-30%, will be counseled on their elevated risk and the option to consider risk-reducing mastectomies as part of their gender-affirming chest masculinization operation. This option will be provided for moderate-risk persons, given the unclear long-term BC risk reduction from chest masculinization surgery alone. Moderate risk individuals will also be counseled on standard risk-reducing strategies, including lifestyle modifications, risk-reducing endocrine therapy options, and increased breast cancer screening strategies.

Participants with a **high lifetime** BC risk, defined as >30%, will be counseled on the potential benefit of undergoing risk-reducing mastectomies as part of their gender-affirming chest masculinization operation, an also be counseled on standard risk-reducing strategies, including lifestyle modifications, risk-reducing endocrine therapy options, and increased breast cancer screening strategies.

Those participants with an elevated lifetime risk based on family history, or with an unknown family history (per NCCN guidelines) will be offered to meet with a Genetic counselor to consider genetic study (see <a href="Section 6.3">Section 6.3</a>).

Those with a moderate or high risk and/or family history suggestive of pathogenic variant who decline further genetic testing or a 2<sup>nd</sup> visit with Dr. Cortina will be given the opportunity to express why they declined.

#### 6.3 Breast Cancer Genetic Testing

Study participants with a family history suggestive of a pathogenic variant and/or with an elevated BC risk who meet NCCN genetic testing guidelines (<u>Appendix 2</u>)<sup>1, 2</sup> will be referred to the Cancer Genetics Clinic to undergo a formal genetic counseling session and possible germline genetic testing. Genetic testing will be performed via the Ambry Genetics<sup>®</sup> Panel, which is our current institution standard.

Persons who undergo genetic testing and are found to have a pathogenic variant for BC will be offered to see the PI, Chandler Cortina, MD, to discuss the utility of risk-reducing mastectomies as part of their chest masculinization operation (see Visit 2). Persons who are found to have a pathogenic variant that infers any other risk besides BC will be referred to the appropriate care teams for further evaluation, as is the current standard practice in our Genetics clinic.


#### 6.4 Visit 2: Surgical Risk-Reducing Mastectomy Counseling

Participants considering risk-reducing mastectomies will meet directly with Dr. Cortina who can perform the operation in tandem with the patient's respective plastic surgeon. Patients who decline risk-reducing mastectomy as part of their surgery will be given the opportunity to express why they declined. This procedure is consistent with the current clinical workflow for cisgender patients. If patients undergo risk-reducing mastectomy as part of their chest masculinization surgery, pathological tissue examination is standard and findings will be collected during the study period.

#### 6.5 Data Factors

Data factors to be collected from study participants for analysis described in <u>Section 9.2.2</u> include the following:

- Name
- DOB
- MRN
- Age
- Weight (lbs)
- Height (inches)
- BMI
- Race
- Ethnicity
- Highest Level of Education
- Insured?
  - o If so, type
- Sex Assigned at Birth
- Gender Identity
- Gender Expression
- Sexual Identity
- History of Gender Affirming Hormone Therapy
  - Duration
  - Dosage
  - Laboratory Values (estrogen, progesterone, and testosterone history)
- Prior Gender-Affirming Surgeries
- Age at First Menstrual Period
- · Age at First Live Birth
  - Number of Children
- Family History Status Known or Unknown?
  - O Unknown Maternal, Paternal, or Both Sides?
- Number of 1<sup>st</sup> Degree Relatives with BC
- Number of 2<sup>nd</sup> Degree Relatives with BC
- Number of 1<sup>st</sup> Degree Relatives with Ovarian Cancer
- Number of 2<sup>nd</sup> Degree Relatives with Ovarian Cancer
- Any Other 1<sup>st</sup> or 2<sup>nd</sup> Degree Relatives with Any Cancer Diagnosis and What Type
- Previous Breast Biopsy

- o If Yes, Atypical Cells
- o If Yes, Pathology
- Any History of Hormone Replacement Therapy (Not Including Gender-affirming Testosterone Therapy)
- Any Ashkenazi Jewish Inheritance?
- Date of Risk Estimation
- Participant's Personal Estimation of Lifetime Risk
- Gail Model Risk Estimate
- IBIS Model Risk Estimate
- Average Risk ([Gail + IBIS Risks]/2)
- Recommended to Undergo Risk-reducing Mastectomies as Part of Top Surgery (Risk 17-30%) (Y/N)
- Given the Option to Consider Risk-reducing Mastectomies as Part of Top Surgery (Risk 17-30%) (Y/N)
- Say they would choose to Undergo Top Surgery (Y/N)
- Underwent Top Surgery (Y/N)
- Underwent Risk-reducing Mastectomies as Part of Top Surgery (Y/N)
- Recommended to Undergo Genetic Counseling (Y/N)
- Underwent Genetic Counseling (Y/N)
- Recommend to Undergo Genetic Testing (Y/N)
- Underwent Genetic Testing (Y/N)
  - o If yes, results:

# 7.0 SUBJECT WITHDRAWAL, END OF STUDY, AND STUDY DISCONTINUATION

#### 7.1 Subject Withdrawal

#### 7.1.1 Patient-Initiated Withdrawal

A participant may decide to withdraw from the study at any time.

#### 7.1.2 Investigator-Initiated Withdrawal

The investigator may withdraw a participant whenever continued participation is no longer in their best interests. Reasons for withdrawing a participant include, but are not limited to, a subject's request to end participation, a subject's noncompliance, or simply significant uncertainty on the part of the investigator that continued participation is prudent.

#### 7.1.3 Replacement Policy and Data Usage

Subjects who sign the informed consent form and are enrolled, but subsequently withdraw, will be replaced. Data collected from subjects that withdraw or discontinue from the study will not be used.

Version No.: 1.0 Version Date: 01/30/23

## 7.2 End of Study Definition

A subject is considered to have completed the study if they have completed all phases of the study including the last scheduled procedure shown in the <u>Study Calendar</u> or has been discontinued.

#### 7.3 Study Discontinuation and Closure

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause (as determined by the MCW study principal investigator, DSMC, sponsor, and/or IRB). Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to study participants, investigator, funding agency, and regulatory authorities. If the study is prematurely terminated or suspended, the MCW principal investigator (PI) will promptly inform the MCW Institutional Review Board (IRB) and sponsor and will provide the reason(s) for the termination or suspension. Study participants will be contacted, as applicable, and be informed of changes.

# 8.0 ADVERSE EVENTS: DEFINITIONS, COLLECTION, AND REPORTING

This study is considered to be of minimal risk to participants due to its design and the nature of the intervention being tested (*i.e.*, risk assessment, genetic testing, and patient education). As described in <u>Section 11.5.1</u>, participants may experience anxiety or distress upon hearing the results of their personalized BC risk assessment and/or their genetic tests.

Subjects will not undergo an investigational medical intervention for the purposes of this study. While the participants' decision to have risk-reducing mastectomies performed in tandem with their gender-affirming chest masculinization procedure will be assessed, the risk-reducing mastectomy procedure itself or its outcomes does not fall under this study protocol. For these reasons, adverse and serious adverse events are not expected, but will be defined, collected, and reported as described in this section if encountered.

#### 8.1 Definitions

#### 8.1.1 Adverse Event (AE)

Any untoward medical occurrence in a subject or clinical investigation subject administered an interventional product and which does not necessarily have to have a causal relationship with this treatment.

This study will utilize the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, located on the CTEP web site:

https://ctep.cancer.gov/protocolDevelopment/electronic applications/ctc.htm

AEs may be spontaneously reported by the subject and/or in response to an open question from study personnel or revealed by observation, physical examination or other diagnostic procedures.


#### 8.1.2 Serious Adverse Event (SAE)

Serious Adverse Event (SAE) means any untoward medical occurrence that results in any of the following outcomes:

- **Death.** Results in death.
- **Life-threatening**. Is life-threatening (refers to an AE in which the participant was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death if it were more severe).
- **Hospitalization**. Requires inpatient hospitalization ≥24 hours or prolongation of an existing hospitalization.
- **Disability/incapacity**. Results in persistent or significant disability or incapacity. (Disability is defined as a substantial disruption of a person's ability to conduct normal life functions).
- Pregnancy
- Medically important event. This refers to an AE that may not result in death, be immediately life threatening, or require hospitalization, but may be considered serious when, based on appropriate medical judgment, may jeopardize the participant, require medical or surgical intervention to prevent one of the outcomes listed above, or involves suspected transmission via a medicinal product of an infectious agent. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse; any organism, virus, or infectious particle (e.g., prion protein transmitting transmissible spongiform encephalopathy), pathogenic or nonpathogenic, is considered an infectious agent.

#### 8.1.3 Attribution of an Adverse Event

An assessment of the relationship between the adverse event and the medical intervention, using the following categories:

- **Definitely Related**: *The AE is clearly related to the intervention*. There is clear evidence to suggest a causal relationship, and other possible contributing factors can be ruled out.
- **Probably Related:** The AE is likely related to the intervention. There is evidence to suggest a causal relationship, and the influence of other factors is unlikely.
- **Possibly Related:** The AE may be related to the intervention. There is some evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time after administration of the trial medication). However, the influence of other factors may have contributed to the event (e.g., the subject's clinical condition, other concomitant events).
- Unlikely: The AE is doubtfully related to the intervention. A clinical event, including an abnormal laboratory test result, whose temporal relationship to drug administration makes a causal relationship improbable (e.g., the event did not occur within a reasonable time after administration of the trial medication) and in which other drugs or chemicals or underlying disease provides plausible explanations (e.g., the subject's clinical condition, other concomitant treatments).

• **Unrelated:** The AE is clearly NOT related to the intervention. The AE is completely independent of study drug administration, and/or evidence exists that the event is definitely related to another etiology.

#### 8.1.4 Expectedness of an Adverse Event

Study Investigator or treating physician will be responsible for determining whether an AE is expected or unexpected as indicated in the protocol, informed consent form and/or drug information brochure. An AE will be considered unexpected if the nature, severity, or frequency of the event is NOT consistent with the risk information previously described for the study intervention.

# 8.2 Collection and Reporting Requirements for Adverse Events and Serious Adverse Events

Adverse and serious adverse events are not expected, but if such events occur, they will be reported per IRB guidelines. Any events reported to the IRB will be reported to the DSMC following the same manner (routine or expedited).

For routine reporting, the events will be reported to the IRB as part of the annual continuing progress report, and the DSMC will review events entered into OnCore<sup>™</sup> at the time of scheduled monitoring.

For expedited DSMC reporting, the study coordinator/research nurse must notify the DSMC via email. For AEs, include the subject ID, date of event, grade, relatedness, expectedness, and a short narrative. For SAEs, DSMC will review the SAE report entered into the secure Microsoft Excel spreadsheet used for the study.

## 8.3 Unanticipated Problem Involving Risk to Subject or Other (UPIRSO)

Unanticipated problems will be submitted to IRB of record and the DSMC, according to local policies and procedures. An unanticipated problem is one that is unexpected, possibly, probably, or definitely related to the research described in the paragraph above, and suggests the research places research participants or others at a greater risk of physical or psychological harm than was previously known or recognized.

Since this is an investigator-initiated study, the principal investigator is responsible for reporting unanticipated problems to any regulatory agency and to the IRB. The study investigators and coordinators follow participants per the schedule of events outlined in the <u>Study Calendar</u> to ensure protocol compliance, participant safety, and quality care. Any unanticipated problems detected will be promptly documented by the study coordinator and submitted to the IRB and DSMC within 5 calendar days of study staff's knowledge. These reviews would pick up any unanticipated negative trends among participants.

#### 8.4 Subject Complaints

If a complaint is received by anyone on the study staff, it will be discussed with the study staff and will be addressed on a case-by-case basis. The PI will be notified of any complaints. Complaints will be reported to the IRB if indicated.

If the subject has questions about his or her rights as a study subject, wants to report any problems or complaints, obtain information about the study or offer input, the subject can call the Medical College of Wisconsin/Froedtert Hospital research subject advocate at 414-955-8844. This information is provided to the subject in their consent.

#### 9.0 STATISTICAL CONSIDERATIONS

#### 9.1 Sample Size Determination and Accrual Estimates

This is a pilot patient outcome study with a sample size of N=35, which would result in a 10% margin of error and a 90% exact confidence interval for a true population proportion of TG men with increased risk of breast cancer (assuming that 4 out of 35 participants will be found to have an elevated BC risk). In the future, enrolling 125 TG individuals would allow investigators to obtain a 90% confidence interval with a margin of error of 5%.

The sample size is also in line with reaching our accrual goal within a one-year period, as it represents one third of the patient population currently seen by our plastic surgeons.

#### 9.2 Analysis Plan

#### 9.2.1 Analysis Population

Data from all participants will be used for endpoint analyses. Data from subjects who withdraw or discontinue will be not used.

#### 9.2.2 Endpoint Analysis

Descriptive statistics will be used to summarize participant characteristics and study outcomes for the above study aims. Median and range will be used for summarizing continuous variables; counts and percentages will be used for categorical variables.

To assess and compare the self-perceived breast cancer risk with calculated risk for third primary endpoint, self-perceived risk will be compared to mean BC calculated risk using the Wilcoxon related sample test. Chi-squared tests will be used to assess patient factors associated with under and overestimating self-perceived risk.

#### 9.3 Missing Data

No major missing data relevant to the primary endpoints are anticipated. Unforeseen missing data, if any, will be addressed in consultation with the study statistician.

# 10.0 DATA AND SAFETY MONITORING PLAN (DSMP)

#### 10.1 Data and Safety Management Overview

The Medical College of Wisconsin (MCW) Data Safety Monitoring Committee (DSMC) and the MCW Institutional Review Board (IRB) will approve protocol-specific DSM plans. A local, investigator-initiated trial will be required to be continuously monitored by the principal investigator of the study with biannual safety and progress reports submitted to the DSMC.

The DSMP for this study will involve the following entities:


#### 10.2 Study Team

The study team minimally consists of 1) the principal investigator, Dr. Chandler Cortina, 2) a nurse practitioner, Anna Purdy, APNP, who is a co-investigator on the study, and 3) the study biostatistician. While subjects are on treatment, the principal investigator will meet periodically with the rest of the study team to review the study status. This review will include but not be limited to reportable SAEs and UPIRSOs and an update of the ongoing study summary that describes study progress in terms of the study schema. The appropriateness of further subject enrollment and the specific intervention for a next subject enrollment is addressed. All meetings including attendance should be documented.

#### 10.3 Quality Assurance

The MCWCC Clinical Trials Office (CTO) provides ongoing quality assurance audits.

This study has been categorized as low risk by the MCW Cancer Center (MCWCC) Scientific Review Committee (SRC) and will be reviewed internally by the MCWCC CTO Quality Assurance Staff according to the MCWCC <u>Data and Safety Monitoring Plan</u> and the current version of the MCWCC CTO SOP, 6.5.2 Internal Quality Assurance Reviews.

#### 10.4 DSMC

The Medical College of Wisconsin Cancer Center places the highest priority on ensuring the safety of subjects participating in clinical trials. Every cancer interventional trial conducted at MCW includes a plan for safety and data monitoring.

More information can be found related to the MCWCC Data and Safety Monitoring Plan at the MCWCC website (Data and Safety Monitoring Plan).

This study will be reviewed by the Medical College of Wisconsin Cancer Center Data and Safety Monitoring Committee (MCWCC DSMC). A summary of the MCWCC DSMC activities are as follows:

- Review the clinical trial for data integrity and safety.
- Review all DSM reports.
- Submit a summary of any recommendations related to study conduct.
- Terminate the study if deemed unsafe for the subject.

A copy of the MCWCC Data and Safety Monitoring Plan and membership roster will be maintained in the study research file and updated as membership changes. The committee will review reports from the study principal investigator twice annually (or more frequently if needed) and provide recommendations on trial continuation, suspension or termination as necessary.

Any available DSMC letters will be submitted to the IRB of record as required.

# 11.0 REGULATORY COMPLIANCE, ETHICS, AND STUDY MANAGEMENT

#### 11.1 Ethical Standard

This study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki as stated in 21 CFR §312.120(c)(4), consistent with GCP and all applicable regulatory requirements.

## 11.2 Regulatory Compliance

This study will be conducted in compliance with:

- The protocol.
- Federal regulations, as applicable, including 21 CFR §50 (Protection of Human Subjects/Informed Consent); 21 CFR §56 (Institutional Review Boards) and §312 (Investigational New Drug Application; and 45 CFR §46 Subparts A (Common Rule), B (Pregnant Women, Human Fetuses and Neonates), C (Prisoners), and D (Children), GCP/ICH guidelines, and all applicable regulatory requirements. The IRB must comply with the regulations in 21 CFR §56 and applicable regulatory requirements.

#### 11.3 Informed Consent Process

Informed consent is a process that is initiated prior to the individual agreeing to participate in the study and continues throughout the individual's study participation. Discussion of the risks and possible benefits of this study will be provided to subjects and their families. Consent forms describing in detail the study objectives, procedures, and risks are given to the subject and documentation of informed consent is required prior to enrollment. Consent forms will include the MCW IRB template language and must be approved by the MCW IRB.

The patient will be asked to read and review the document. Upon reviewing the document, the investigators will explain the research study to the patient and answer any questions that may arise. In accordance with 46 CFR §46.111, the patient will sign and date the informed consent document prior to any procedures being done specifically for the study. A witness should only sign when required, per FH/MCW IRB policy. The subjects will have the opportunity to discuss the study with their surrogates or think about it prior to agreeing to participate. The subjects may withdraw consent at any time throughout the course of the trial.

If the patient signs the consent form, the original signed document will become part of the patient's medical records and the patient will receive a copy of the signed document.

## 11.4 Subject Confidentiality and Access to Source Documents/Data

Subject confidentiality is strictly held in trust by the principal investigator, participating investigators, and any staff. This confidentiality includes the clinical information relating to participating subjects, as well as any genetic or biological testing.

The study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or data will be released to any unauthorized third party without prior written approval of the principal investigator. The conditions for maintaining

confidentiality of the subjects' records are required for the life of the data. These rules apply equally to any and all MCWCC projects.

The principal investigator will allow access to all source data and documents for the purposes of monitoring, audits, IRB review and regulatory inspections.

The study monitor or other authorized representatives of the principal investigator may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the subjects in this study. The clinical study site will permit access to such records.

#### 11.5 Risk-Benefit Assessment

#### 11.5.1 Potential and Protections Against Risks

There is the potential for participant anxiety or distress regarding the results of their personalized BC risk assessment and/or their genetic test results. Our study team will do our best to answer questions and assuage concerns regarding anxiety of distress of testing results, we are also supported by the psychiatry and social work teams in the Clinical Cancer Center.

Another risk of taking part in a research study is that more people will handle the personal health information collected for this study. The study team will make every effort to protect the information and keep it confidential (see <u>Section 10.1</u>), but it is possible that an unauthorized person might see it. Depending on the kind of information being collected, it might be used in a way that could embarrass the subject or affect his/her ability to get insurance.

#### 11.5.2 Potential Benefits

Participants will be informed of their personal breast cancer risk which may influence if they undergo top surgery and how they undergo top surgery. This may also influence if they should consider genetic testing which may also impact their family members.

Findings from this proposal will inform the TGNB community and healthcare providers on how instituting a personalized BC risk assessment impacts surgical-decision regarding chest masculinization surgery.

For these reasons, the potential benefits of the study are reasonable in relation to the anticipated risks to the study participants.

#### 11.6 Protection of Human Subjects

#### 11.6.1 Protection from Unnecessary Harm

Each clinical site is responsible for protecting all subjects involved in human experimentation. This is accomplished through the IRB mechanism and the informed consent process. The IRB reviews all proposed studies involving human experimentation and ensures that the subject's rights and welfare are protected and that the potential benefits and/or the importance of the knowledge to be gained outweigh the risks to the individual. The IRB also reviews the informed consent document associated with each study in order to ensure that the consent document accurately and clearly communicates the nature of the research to be done and its associated risks and benefits.

#### 11.6.2 Protection of Privacy

To ensure confidentiality, each participant is assigned an anonymous study ID, which is then used on all study forms that collect participant data. Study IDs are linked to participant names and other private identifiable information in only one location, on an encrypted, firewall protected, electronic document housed on MCW's server. All study forms are to be kept on an MCW password-protected computer, server, or HIPAA compliant data sharing platform, with access restricted to authorized study personnel.

#### 11.7 Changes in the Protocol

Once the protocol has been approved by the MCW IRB, any changes to the protocol must be documented in the form of an amendment. The amendment must be signed by the investigator and approved by the IRB prior to implementation.

If it becomes necessary to alter the protocol to eliminate an immediate hazard to subjects, an amendment may be implemented prior to IRB approval. In this circumstance, however, the investigator must then notify the IRB in writing within five working days after implementation.

The IRB may provide, if applicable regulatory authority(ies) permit, expedited review and approval/favorable opinion for minor change(s) in ongoing studies that have the approval /favorable opinion of the IRB. The investigator will submit all protocol modifications to the sponsor and the regulatory authority(ies) in accordance with the governing regulations.

Changes to the protocol may require approval from the sponsor.

Any deviations from the protocol must be fully documented in the source documents and reported to the IRB per institutional guidelines.

#### 11.8 Investigator Compliance

The investigator will conduct the study in compliance with the protocol given approval/favorable opinion by the IRB and the appropriate regulatory authority(ies).

Onsite Audits: Auditing is essential to ensure that research conducted at the Medical College of Wisconsin (MCW) Cancer Center is of the highest quality and meets MCW and regulatory agency standards.

Regulatory authorities, the IRB, and/or sponsor may request access to all source documents, data capture records and other study documentation for onsite audit or inspection. Direct access to these documents must be guaranteed by the investigator, who must provide support at all times for these activities.

The PI will follow the procedures as outlined above, which will serve as part of the quality control procedure. The PI will also meet with the mentorship team and CRC regularly to ensure data accuracy, appropriate data analysis, and protocol adherence. To ensure the validity and integrity of study data, the PI will discuss data management with the research team and CRC on a regular basis.

#### 12.0 DATA MANAGEMENT

#### 12.1 Data Management Plan

Study electronic data will be stored on a password-protected Microsoft Excel file using password-protected computers on encrypted networks that are backed up nightly. In addition to protected health information (PHI) data (name, date of birth and medical record number), other data to be collected include participant demographic information (race, ethnicity, age, sex assigned at birth, gender, etc.), initial VAS personal estimate, results from the personalized BC risk assessment, possible genetic testing results, and the type of gender-affirming chest masculinization surgery the participant undergoes. Initial intake data will be entered into Qualtrics, a secure online survey platform, at the time of personalized BC risk assessment, and then converted to a Microsoft Excel file where subsequent patient data (genetic test results, decision for surgery) will be directly entered by the PI and Co-I. All data will be de-identified prior to statistical analysis. All consent forms will be kept in locked file cabinets in locked offices.

#### 12.2 Disseminating and Publishing Data

All raw data, data figures, data interpretation, models, and conclusions drawn from this study will be managed by the principal investigator and co-investigators listed in this protocol. The findings from this study may be presented at relevant conferences/meetings, published in a respectable peer-reviewed journal, or used as preliminary data in a grant application to justify extramural funding.

For any manuscript that is to be published in a journal, the role of authors/contributors, the disclosure of financial/non-financial relationships and activities, and the report of perceived conflicts of interest will largely adhere to the recommended guidelines set forth by the International Committee of Medical Journal Editors (ICMJE; Defining the Role of Authors and Contributors, Disclosure of Financial and Non-Financial Relationship and Activities and Conflicts of Interest). The PI, in consultation with the study co-investigators, will determine who will be listed as first, senior, and corresponding author(s). Study team members who have made substantial and significant intellectual contributions to the study and its findings will be listed as contributing authors or, in certain circumstances, acknowledged. Funding sources and any conflict of interests, perceived or actual, will be disclosed and stated within the appropriate section of the manuscript at submission.


#### REFERENCES

- Manahan ER, Kuerer HM, Sebastian M, Hughes KS, Boughey JC, Euhus DM, Boolbol SK, Taylor WA. Consensus Guidelines on Genetic` Testing for Hereditary Breast Cancer from the American Society of Breast Surgeons. Annals of Surgical Oncology. 2019;26(10):3025-31. doi: 10.1245/s10434-019-07549-8.
- Daly MB, Pal T, Berry MP, Buys SS, Dickson P, Domchek SM, Elkhanany A, Friedman S, Goggins M, Hutton ML, CGC, Karlan BY, Khan S, Klein C, Kohlmann W, CGC, Kurian AW, Laronga C, Litton JK, Mak JS, LCGC, Menendez CS, Merajver SD, Norquist BS, Offit K, Pederson HJ, Reiser G, CGC, Senter-Jamieson L, CGC, Shannon KM, Shatsky R, Visvanathan K, Weitzel JN, Wick MJ, Wisinski KB, Yurgelun MB, Darlow SD, Dwyer MA. Genetic/Familial High-Risk Assessment: Breast, Ovarian, and Pancreatic, Version 2.2021, NCCN Clinical Practice Guidelines in Oncology. Journal of the National Comprehensive Cancer Network. 2021;19(1):77-102. doi: 10.6004/jnccn.2021.0001.
- 3. Canner JK, Harfouch O, Kodadek LM, Pelaez D, Coon D, Offodile AC, II, Haider AH, Lau BD. Temporal Trends in Gender-Affirming Surgery Among Transgender Patients in the United States. JAMA Surgery. 2018;153(7):609-16. doi: 10.1001/jamasurg.2017.6231.
- 4. About 5% of young adults in the U.S. say their gender is different from their sex assigned at birth: Pew Research Center; 2022 [updated June 7, 2022]. Available from: <a href="https://www.pewresearch.org/fact-tank/2022/06/07/about-5-of-young-adults-in-the-u-s-say-their-gender-is-different-from-their-sex-assigned-at-birth/">https://www.pewresearch.org/fact-tank/2022/06/07/about-5-of-young-adults-in-the-u-s-say-their-gender-is-different-from-their-sex-assigned-at-birth/</a>.
- 5. Meerwijk EL, Sevelius JM. Transgender Population Size in the United States: a Meta-Regression of Population-Based Probability Samples. American Journal of Public Health. 2017;107(2):e1-e8. doi: 10.2105/ajph.2016.303578. PubMed PMID: 28075632.
- 6. Akhavan AA, Sandhu S, Ndem I, Ogunleye AA. A review of gender affirmation surgery: What we know, and what we need to know. Surgery. 2021;170(1):336-40. doi: https://doi.org/10.1016/j.surg.2021.02.013.
- Clarke CN, Cortina CS, Fayanju OM, Dossett LA, Johnston FM, Wong SL. Breast Cancer Risk and Screening in Transgender Persons: A Call for Inclusive Care. Annals of Surgical Oncology. 2022;29(4):2176-80. doi: 10.1245/s10434-021-10217-5.
- 8. Jatoi I, Kemp Z. Risk-Reducing Mastectomy. JAMA. 2021;325(17):1781-2. doi: 10.1001/jama.2020.22414.
- 9. Jakub JW, Peled AW, Gray RJ, Greenup RA, Kiluk JV, Sacchini V, McLaughlin SA, Tchou JC, Vierkant RA, Degnim AC, Willey S. Oncologic Safety of Prophylactic Nipple-Sparing Mastectomy in a Population With BRCA Mutations: A Multi-institutional Study. JAMA Surgery. 2018;153(2):123-9. doi: 10.1001/jamasurg.2017.3422.
- Garstka M, Henriquez A, Kelly BN, Webster A, Khubchandani JA, Hughes K, Nguyen A, Oseni T, Specht M, Coopey SB, Gadd MA, Smith BL. How Protective are Nipple-Sparing Prophylactic Mastectomies in BRCA1 and BRCA2 Mutation Carriers? Annals of Surgical Oncology. 2021;28(10):5657-62. doi: 10.1245/s10434-021-10445-9.
- 11. Stone JP, Hartley RL, Temple-Oberle C. Breast cancer in transgender patients: A systematic review. Part 2: Female to Male. European Journal of Surgical Oncology. 2018;44(10):1463-8. doi: https://doi.org/10.1016/j.ejso.2018.06.021.
- 12. de Blok CJM, Wiepjes CM, Nota NM, van Engelen K, Adank MA, Dreijerink KMA, Barbé E, Konings IRHM, den Heijer M. Breast cancer risk in transgender people receiving hormone treatment: nationwide cohort study in the Netherlands. BMJ. 2019;365:I1652. doi: 10.1136/bmj.I1652.
- 13. Brown GR, Jones KT. Incidence of breast cancer in a cohort of 5,135 transgender veterans. Breast Cancer Research and Treatment. 2015;149(1):191-8. doi: 10.1007/s10549-014-3213-2.

- 14. Cortina CS, Kong AL. Chest Mass in a Transgender Man after Top Surgery. Lancet Oncology.In Press.
- 15. Almazan AN, Keuroghlian AS. Association Between Gender-Affirming Surgeries and Mental Health Outcomes. JAMA Surgery. 2021;156(7):611-8. doi: 10.1001/jamasurg.2021.0952.
- 16. Cortina CS. Inclusion and Reporting of Transgender and Nonbinary Persons in Clinical Trials and Tumor Registries—The Time Is Now. JAMA Oncology. 2022;8(8):1097-8. doi: 10.1001/jamaoncol.2022.1638.
- 17. Safer JD. Research gaps in medical treatment of transgender/nonbinary people. The Journal of Clinical Investigation. 2021;131(4). doi: 10.1172/JCI142029.
- 18. Martinez EO, Rubin M, Miller T, Cortina CS. Transgender and Non-binary Persons in Contemporary Oncology Randomized Clinical Trials. Annals of Surgical Oncology. 2022;29(13):7958-60. doi: 10.1245/s10434-022-12418-y.
- Wetmore JB, Otarola L, Paulino LJ, Henry BR, Levine AF, Kone D, Ulloa J, Jandorf L, Margolies L, Vang S. Estimating lifetime risk for breast cancer as a screening tool for identifying those who would benefit from additional services among women utilizing mobile mammography. Journal of Cancer Policy. 2022;34:100354. doi: <a href="https://doi.org/10.1016/j.jcpo.2022.100354">https://doi.org/10.1016/j.jcpo.2022.100354</a>.
- 20. How common is breast cancer? : American Cancer Society; 2022 [updated October 6, 2022; cited 2022 August 30]. Available from: <a href="https://www.cancer.org/cancer/breast-cancer/about/how-common-is-breast-cancer.html">https://www.cancer.org/cancer/breast-cancer/about/how-common-is-breast-cancer.html</a>.
- 21. King TA, Sakr RA, Muhsen S, Andrade VP, Giri D, Van Zee KJ, Morrow M. Is There a Low-Grade Precursor Pathway in Breast Cancer? Annals of Surgical Oncology. 2012;19(4):1115-21. doi: 10.1245/s10434-011-2053-0.
- 22. King TA, Pilewskie M, Muhsen S, Patil S, Mautner SK, Park A, Oskar S, Guerini-Rocco E, Boafo C, Gooch JC, Brot MD, Reis-Filho JS, Morrogh M, Andrade VP, Sakr RA, Morrow M. Lobular Carcinoma in Situ: A 29-Year Longitudinal Experience Evaluating Clinicopathologic Features and Breast Cancer Risk. Journal of Clinical Oncology. 2015;33(33):3945-52. doi: 10.1200/jco.2015.61.4743. PubMed PMID: 26371145.
- 23. Rageth CJ, Rubenov R, Bronz C, Dietrich D, Tausch C, Rodewald A-K, Varga Z. Atypical ductal hyperplasia and the risk of underestimation: tissue sampling method, multifocality, and associated calcification significantly influence the diagnostic upgrade rate based on subsequent surgical specimens. Breast Cancer. 2019;26(4):452-8. doi: 10.1007/s12282-018-00943-2.
- 24. Moskowitz CS, Ronckers CM, Chou JF, Smith SA, Friedman DN, Barnea D, Kok JL, Vries Sd, Wolden SL, Henderson TO, Pal HJHvd, Kremer LCM, Neglia JP, Turcotte LM, Howell RM, Arnold MA, Schaapveld M, Aleman B, Janus C, Versluys B, Leisenring W, Sklar CA, Begg CB, Pike MC, Armstrong GT, Robison LL, Leeuwen FEv, Oeffinger KC. Development and Validation of a Breast Cancer Risk Prediction Model for Childhood Cancer Survivors Treated With Chest Radiation: A Report From the Childhood Cancer Survivor Study and the Dutch Hodgkin Late Effects and LATER Cohorts. Journal of Clinical Oncology. 2021;39(27):3012-21. doi: 10.1200/jco.20.02244. PubMed PMID: 34048292.
- 25. Canet M, Harbron R, Thierry-Chef I, Cardis E. Cancer Effects of Low to Moderate Doses of Ionizing Radiation in Young People with Cancer-Predisposing Conditions: A Systematic Review. Cancer Epidemiology, Biomarkers & Prevention. 2022;31(10):1871-89. doi: 10.1158/1055-9965.Epi-22-0393.
- 26. Kuchenbaecker KB, Hopper JL, Barnes DR, Phillips K-A, Mooij TM, Roos-Blom M-J, Jervis S, van Leeuwen FE, Milne RL, Andrieu N, Goldgar DE, Terry MB, Rookus MA, Easton DF, Antoniou AC, BRCA1 at, Consortium BC. Risks of Breast, Ovarian, and Contralateral Breast Cancer for BRCA1 and BRCA2 Mutation Carriers. JAMA. 2017;317(23):2402-16. doi: 10.1001/jama.2017.7112.

- 27. Baxter JS, Leavy OC, Dryden NH, Maguire S, Johnson N, Fedele V, Simigdala N, Martin L-A, Andrews S, Wingett SW, Assiotis I, Fenwick K, Chauhan R, Rust AG, Orr N, Dudbridge F, Haider S, Fletcher O. Capture Hi-C identifies putative target genes at 33 breast cancer risk loci. Nature Communications. 2018;9(1):1028. doi: 10.1038/s41467-018-03411-9.
- 28. Veitinger JK, Kerber AS, Gabram-Mendola SGA, Liu Y, Durham LM, Durrence D, Berzen AK, Shin JY, Snyder C, Bellcross CA, Guan Y. Screening for Individuals at Risk for Hereditary Breast and Ovarian Cancer: A Statewide Initiative, Georgia, 2012–2020. American Journal of Public Health. 2022;112(9):1249-52. doi: 10.2105/ajph.2022.306932. PubMed PMID: 35862880.
- 29. Maas P, Barrdahl M, Joshi AD, Auer PL, Gaudet MM, Milne RL, Schumacher FR, Anderson WF, Check D, Chattopadhyay S, Baglietto L, Berg CD, Chanock SJ, Cox DG, Figueroa JD, Gail MH, Graubard BI, Haiman CA, Hankinson SE, Hoover RN, Isaacs C, Kolonel LN, Le Marchand L, Lee I-M, Lindström S, Overvad K, Romieu I, Sanchez M-J, Southey MC, Stram DO, Tumino R, VanderWeele TJ, Willett WC, Zhang S, Buring JE, Canzian F, Gapstur SM, Henderson BE, Hunter DJ, Giles GG, Prentice RL, Ziegler RG, Kraft P, Garcia-Closas M, Chatterjee N. Breast Cancer Risk From Modifiable and Nonmodifiable Risk Factors Among White Women in the United States. JAMA Oncology. 2016;2(10):1295-302. doi: 10.1001/jamaoncol.2016.1025.
- 30. Shin YE, Gail MH, Pfeiffer RM. Assessing risk model calibration with missing covariates. Biostatistics. 2021;23(3):875-90. doi: 10.1093/biostatistics/kxaa060.
- 31. Rockhill B, Spiegelman D, Byrne C, Hunter DJ, Colditz GA. Validation of the Gail et al. Model of Breast Cancer Risk Prediction and Implications for Chemoprevention. JNCI: Journal of the National Cancer Institute. 2001;93(5):358-66. doi: 10.1093/jnci/93.5.358.
- 32. Chay WY, Ong WS, Tan PH, Jie Leo NQ, Ho GH, Wong CS, Chia KS, Chow KY, Tan M, Ang P. Validation of the Gail model for predicting individual breast cancer risk in a prospective nationwide study of 28,104 Singapore women. Breast Cancer Research. 2012;14(1):R19. doi: 10.1186/bcr3104.
- 33. Nickson C, Procopio P, Velentzis LS, Carr S, Devereux L, Mann GB, James P, Lee G, Wellard C, Campbell I. Prospective validation of the NCI Breast Cancer Risk Assessment Tool (Gail Model) on 40,000 Australian women. Breast Cancer Research. 2018;20(1):155. doi: 10.1186/s13058-018-1084-x.
- 34. Stark GF, Hart GR, Nartowt BJ, Deng J. Predicting breast cancer risk using personal health data and machine learning models. PLOS ONE. 2019;14(12):e0226765. doi: 10.1371/journal.pone.0226765.
- 35. Gail MH, Mai PL. Comparing Breast Cancer Risk Assessment Models. JNCI: Journal of the National Cancer Institute. 2010;102(10):665-8. doi: 10.1093/jnci/djq141.
- 36. Pal Choudhury P, Wilcox AN, Brook MN, Zhang Y, Ahearn T, Orr N, Coulson P, Schoemaker MJ, Jones ME, Gail MH, Swerdlow AJ, Chatterjee N, Garcia-Closas M. Comparative Validation of Breast Cancer Risk Prediction Models and Projections for Future Risk Stratification. JNCI: Journal of the National Cancer Institute. 2019;112(3):278-85. doi: 10.1093/jnci/djz113.
- 37. Kurian AW, Hughes E, Simmons T, Bernhisel R, Probst B, Meek S, Caswell-Jin JL, John EM, Lanchbury JS, Slavin TP, Wagner S, Gutin A, Rohan TE, Shadyab AH, Manson JE, Lane D, Chlebowski RT, Stefanick ML. Performance of the IBIS/Tyrer-Cuzick model of breast cancer risk by race and ethnicity in the Women's Health Initiative. Cancer. 2021;127(20):3742-50. doi: <a href="https://doi.org/10.1002/cncr.33767">https://doi.org/10.1002/cncr.33767</a>.
- 38. Valero MG, Zabor EC, Park A, Gilbert E, Newman A, King TA, Pilewskie ML. The Tyrer–Cuzick Model Inaccurately Predicts Invasive Breast Cancer Risk in Women With LCIS. Annals of Surgical Oncology. 2020;27(3):736-40. doi: 10.1245/s10434-019-07814-w.
- 39. Gallagher S, Hughes E, Kurian AW, Domchek SM, Garber J, Probst B, Morris B, Tshiaba P, Meek S, Rosenthal E, Roa B, Slavin TP, Wagner S, Weitzel J, Gutin A, Lanchbury JS,

- Robson M. Comprehensive Breast Cancer Risk Assessment for CHEK2 and ATM Pathogenic Variant Carriers Incorporating a Polygenic Risk Score and the Tyrer-Cuzick Model. JCO Precision Oncology. 2021(5):1073-81. doi: 10.1200/po.20.00484.
- 40. Stevanato KP, Pedroso RB, Iora P, Santos Ld, Pelloso FC, Melo WAd, Carvalho MDdB, Pelloso SM. Comparative Analysis between the Gail, Tyrer-Cuzick and BRCAPRO Models for Breast Cancer Screening in Brazilian Population. Asian Pacific Journal of Cancer Prevention. 2019;20(11):3407-13. doi: 10.31557/apjcp.2019.20.11.3407.
- 41. Brentnall AR, Cuzick J. Risk Models for Breast Cancer and Their Validation. Statistical Science. 2020;35(1):14-30, 17.
- 42. Brentnall AR, Cuzick J, Buist DSM, Bowles EJA. Long-term Accuracy of Breast Cancer Risk Assessment Combining Classic Risk Factors and Breast Density. JAMA Oncology. 2018;4(9):e180174-e. doi: 10.1001/jamaoncol.2018.0174.
- 43. Hughes E, Tshiaba P, Wagner S, Judkins T, Rosenthal E, Roa B, Gallagher S, Meek S, Dalton K, Hedegard W, Adami CA, Grear DF, Domchek SM, Garber J, Lancaster JM, Weitzel JN, Kurian AW, Lanchbury JS, Gutin A, Robson ME. Integrating Clinical and Polygenic Factors to Predict Breast Cancer Risk in Women Undergoing Genetic Testing. JCO Precision Oncology. 2021(5):307-16. doi: 10.1200/po.20.00246.
- 44. National Collaborating Centre for C. Familial Breast Cancer: Classification and Care of People at Risk of Familial Breast Cancer and Management of Breast Cancer and Related Risks in People with a Family History of Breast Cancer. National Collaborating Centre for Cancer (UK), Cardiff (UK); 2013.
- 45. Understanding Risk: Susan G. Komen 2022 [updated April 29, 2022; cited 2022 August 30]. Available from: <a href="https://www.komen.org/breast-cancer/risk-factor/understanding-risks/">https://www.komen.org/breast-cancer/risk-factor/understanding-risks/</a>.
- 46. DeCensi A, Puntoni M, Guerrieri-Gonzaga A, Caviglia S, Avino F, Cortesi L, Taverniti C, Pacquola MG, Falcini F, Gulisano M, Digennaro M, Cariello A, Cagossi K, Pinotti G, Lazzeroni M, Serrano D, Branchi D, Campora S, Petrera M, Webber TB, Boni L, Bonanni B. Randomized Placebo Controlled Trial of Low-Dose Tamoxifen to Prevent Local and Contralateral Recurrence in Breast Intraepithelial Neoplasia. Journal of Clinical Oncology. 2019;37(19):1629-37. doi: 10.1200/jco.18.01779. PubMed PMID: 30973790.
- 47. Monticciolo DL, Newell MS, Moy L, Niell B, Monsees B, Sickles EA. Breast Cancer Screening in Women at Higher-Than-Average Risk: Recommendations From the ACR. Journal of the American College of Radiology. 2018;15(3, Part A):408-14. doi: https://doi.org/10.1016/j.jacr.2017.11.034.
- 48. Mariscotti G, Belli P, Bernardi D, Brancato B, Calabrese M, Carbonaro LA, Cavallo-Marincola B, Caumo F, Clauser P, Martinchich L, Montemezzi S, Panizza P, Pediconi F, Tagliafico A, Trimboli RM, Zuiani C, Sardanelli F. Mammography and MRI for screening women who underwent chest radiation therapy (lymphoma survivors): recommendations for surveillance from the Italian College of Breast Radiologists by SIRM. La radiologia medica. 2016;121(11):834-7. doi: 10.1007/s11547-016-0667-9.
- 49. Provinciali N, Suen C, Dunn BK, DeCensi A. Raloxifene hydrochloride for breast cancer risk reduction in postmenopausal women. Expert Review of Clinical Pharmacology. 2016;9(10):1263-72. doi: 10.1080/17512433.2016.1231575.
- 50. Heemskerk-Gerritsen BAM, Jager A, Koppert LB, Obdeijn AI-M, Collée M, Meijers-Heijboer HEJ, Jenner DJ, Oldenburg HSA, van Engelen K, de Vries J, van Asperen CJ, Devilee P, Blok MJ, Kets CM, Ausems MGEM, Seynaeve C, Rookus MA, Hooning MJ. Survival after bilateral risk-reducing mastectomy in healthy BRCA1 and BRCA2 mutation carriers. Breast Cancer Research and Treatment. 2019;177(3):723-33. doi: 10.1007/s10549-019-05345-2.
- 51. Tung NM, Boughey JC, Pierce LJ, Robson ME, Bedrosian I, Dietz JR, Dragun A, Gelpi JB, Hofstatter EW, Isaacs CJ, Jatoi I, Kennedy E, Litton JK, Mayr NA, Qamar RD, Trombetta MG, Harvey BE, Somerfield MR, Zakalik D. Management of Hereditary Breast Cancer: American Society of Clinical Oncology, American Society for Radiation Oncology, and

- Society of Surgical Oncology Guideline. Journal of Clinical Oncology. 2020;38(18):2080-106. doi: 10.1200/jco.20.00299. PubMed PMID: 32243226.
- 52. Domchek SM, Friebel TM, Singer CF, Evans DG, Lynch HT, Isaacs C, Garber JE, Neuhausen SL, Matloff E, Eeles R, Pichert G, Van t'veer L, Tung N, Weitzel JN, Couch FJ, Rubinstein WS, Ganz PA, Daly MB, Olopade OI, Tomlinson G, Schildkraut J, Blum JL, Rebbeck TR. Association of Risk-Reducing Surgery in BRCA1 or BRCA2 Mutation Carriers With Cancer Risk and Mortality. JAMA. 2010;304(9):967-75. doi: 10.1001/jama.2010.1237.
- 53. Schultz KAP, Rednam SP, Kamihara J, Doros L, Achatz MI, Wasserman JD, Diller LR, Brugières L, Druker H, Schneider KA, McGee RB, Foulkes WD. PTEN, DICER1, FH, and Their Associated Tumor Susceptibility Syndromes: Clinical Features, Genetics, and Surveillance Recommendations in Childhood. Clinical Cancer Research. 2017;23(12):e76-e82. doi: 10.1158/1078-0432.Ccr-17-0629.
- 54. Corso G, Intra M, Trentin C, Veronesi P, Galimberti V. CDH1 germline mutations and hereditary lobular breast cancer. Familial Cancer. 2016;15(2):215-9. doi: 10.1007/s10689-016-9869-5.
- 55. Antoniou AC, Casadei S, Heikkinen T, Barrowdale D, Pylkäs K, Roberts J, Lee A, Subramanian D, De Leeneer K, Fostira F, Tomiak E, Neuhausen SL, Teo ZL, Khan S, Aittomäki K, Moilanen JS, Turnbull C, Seal S, Mannermaa A, Kallioniemi A, Lindeman GJ, Buys SS, Andrulis IL, Radice P, Tondini C, Manoukian S, Toland AE, Miron P, Weitzel JN, Domchek SM, Poppe B, Claes KBM, Yannoukakos D, Concannon P, Bernstein JL, James PA, Easton DF, Goldgar DE, Hopper JL, Rahman N, Peterlongo P, Nevanlinna H, King M-C, Couch FJ, Southey MC, Winqvist R, Foulkes WD, Tischkowitz M. Breast-Cancer Risk in Families with Mutations in PALB2. New England Journal of Medicine. 2014;371(6):497-506. doi: 10.1056/NEJMoa1400382. PubMed PMID: 25099575.
- 56. Roeb W, Higgins J, King M-C. Response to DNA damage of CHEK2 missense mutations in familial breast cancer. Human Molecular Genetics. 2012;21(12):2738-44. doi: 10.1093/hmg/dds101.
- 57. Cragun D, Weidner A, Tezak A, Clouse K, Pal T. Cancer risk management among female BRCA1/2, PALB2, CHEK2, and ATM carriers. Breast Cancer Research and Treatment. 2020;182(2):421-8. doi: 10.1007/s10549-020-05699-y.
- 58. Carbine NE, Lostumbo L, Wallace J, Ko H. Risk-reducing mastectomy for the prevention of primary breast cancer. Cochrane Database of Systematic Reviews. 2018(4). doi: 10.1002/14651858.CD002748.pub4. PubMed PMID: CD002748.
- 59. Bedrosian I, Parker PA, Brewster AM. Who should get a contralateral prophylactic mastectomy for breast cancer? Cancer. 2019;125(9):1400-3. doi: https://doi.org/10.1002/cncr.31915.
- 60. Hajian-Tilaki K, Nikpour M. Accuracy of self-perceived risk perception of breast cancer development in Iranian women. BMC Women's Health. 2021;21(1):93. doi: 10.1186/s12905-021-01238-z.
- 61. de Jonge ET, Vlasselaer J, Van de Putte G, Schobbens JC. The construct of breast cancer risk perception: need for a better risk communication? Facts Views Vis Obgyn. 2009;1(2):122-9. Epub 2009/01/01. PubMed PMID: 25478077; PMCID: PMC4251271.
- 62. Fehniger J, Livaudais-Toman J, Karliner L, Kerlikowske K, Tice JA, Quinn J, Ozanne E, Kaplan CP. Perceived versus objective breast cancer risk in diverse women. J Womens Health (Larchmt). 2014;23(5):420-7. Epub 2014/01/01. doi: 10.1089/jwh.2013.4516. PubMed PMID: 24372085; PMCID: PMC4011422.
- 63. Cortina CS. Assessing Breast and Ovarian Cancer Risk Prior To Gender-Affirming Surgery. JAMA Surgery.In Press.

# APPENDIX 1. LIFETIME BREAST CANCER RISK ASSESSMENT FORM

#### **Lifetime Breast Cancer Risk Estimation**

| Name: | | | | | |
|---|---|---|---|---|---|
| Date:/2022 | | | | | |
| Participant reported lifetime risk estimation | on:% | | | | |
| 0 10 20 30 40 | 11111111111111111111111111111111111111 | 70 | 1111111111<br>80 | 11 111 11<br>90 | Щ<br>100 |
| Green arrow depicts is the average lifetime risk for cisgender women up to age 85. | | | | | |
| Gail model reported lifetime risk estimation | on (for those 35 and | d older): | % | | |
| IBIS model lifetime risk estimation: | % | | | | |



Gail Model: https://www.mdcalc.com/calc/3647/gail-model-breast-cancer-risk

IBIS Model: https://ibis.ikonopedia.com


## APPENDIX 2. NCCN TESTING CRITERIA FOR HIGH-PENETRANCE BREAST AND/OR OVARIAN CANCER SUSCEPTIBILITY GENES

TESTING CRITERIA FOR HIGH-PENETRANCE BREAST AND/OR OVARIAN CANCER SUSCEPTIBILITY GENES (This can include *BRCA1*, *BRCA2*, *CDH1*, *PALB2*, *PTEN*, and *TP53* among others. See GENE-A for a more complete list.)<sup>a,b,c,d</sup> Testing is clinically indicated in the following scenarios: 1. Individuals with any blood relative with a known pathogenic/likely pathogenic variant in a cancer susceptibility gene
2. Individuals meeting the criteria below but tested negative with previous limited testing (eg, single gene and/or absent deletion duplication analysis) interested in pursuing multi-gene testing absent deletion duplication analysis) interested in pursuing multi-gene testing

3. Personal history of cancer

Breast cancer with at least one of the following:

Diagnosed at age ≤45 y; or

Diagnosed at age 46–50 y with:

Unknown or limited family history; or

A second breast cancer diagnosed at any age; or

≥1 close blood relative! with breast, ovarian, pancreatic, or prostate cancer at any age

Diagnosed at age ≤60 y with triple-negative breast cancer;

Diagnosed at any age with:

Ashkenazi Jewish ancestry; or

≥1 close blood relative! with breast cancer at age ≤50 y or ovarian, pancreatic, metastatic, intraductal/ cribriform histology, or high- or very-high risk group (see NCCN Guidelines for Prostate Cancer) prostate cancer at any age; or Criteria → See GENE-1\* met If criteria If testing for other cancer at any age; or hereditary ♦ ≥3 total diagnoses of breast cancer in patient and/or close blood relatives criteria not met. syndromes Diagnosed at any age with male breast cancer
 Epithelial ovarian cancer<sup>h</sup> (including fallopian tube cancer or peritoneal cancer) at any age consider not met, Exocrine pancreatic cancer at any age (See CRIT-3\*) testina then cancer · Prostate cancer at any age with: for other screening ▶ Metastatic,<sup>g</sup> intraductal/cribriform histology, or high- or very-high-risk group (see NCCN Guidelines for Prostate hereditary syndromes NCCN Any NCCN risk group (see NCCN Guidelines for Prostate Cancer) with the following family history: Screening ♦ Ashkenazi Jewish ancestry; or
 ♦≥1 close relative with breast cancer at age ≤50 y or ovarian, pancreatic, metastatic,<sup>9</sup> or intraductal/cribriform Guidelines† or Close relative with bleast cancer at age 250 y or ovariant, parior cardy, included, included prostate cancer at any age; or 

or ≥2 close relatives with either breast or prostate cancer (any grade) at any age

• A mutation identified on tumor genomic testing that has clinical implications if also identified in the germline

• Individual who meets Li-Fraumeni syndrome (LFS) testing criteria (see CRIT-4\*) or Cowden syndrome/PTEN **Footnotes** on CRIT-2A\* \*To aid in systemic therapy decision-making, such as for HER2-negative metastatic breast cancer Continued on next page \*Available online, in these guidelines, at NCCN.org. †To view the most recent version of these guidelines, visit NCCN.org. Version 2,2021, 11/20/20 © National Comprehensive Cancer Network, Inc. 2021. All rights reserved.

The NCCN Guidelines® and this illustration may not be reproduced in any form without the express written permission of NCCN. CRIT-1 TESTING CRITERIA FOR HIGH-PENETRANCE BREAST AND/OR OVARIAN CANCER SUSCEPTIBILITY GENES (This can include BRCA1, BRCA2, CDH1, PALB2, PTEN, and TP53 among others. See GENE-A for a more complete list.)a,b,c,d Testing is clinically indicated in the following scenarios (continued): Iesting is clinically indicated in the following scenarios (continued):

4. Family history of cancer

• An affected or unaffected individual with a first- or second-degree blood relative meeting any of the criteria listed above (except individuals who meet criteria only for systemic therapy decision-making).

If the affected relative has pancreatic cancer or prostate cancer (metastatic, intraductal/cribriform, or NCCN Guidelines for Prostate Cancer - High- or Very-High-Risk Group), only first-degree relatives should be offered testing unless indicated for other relatives based on additional family history.

• An affected or unaffected individual who otherwise does not meet the criteria above but has a probability >5% of a BRCA1/2 pathogenic variant based on prior probability models (eg, Tyrer-Cuzick, BRCAPro, CanRisk) Criteria → See GENE-1\* met Testing may be considered in the following scenarios (with appropriate pre-test education and access to post-test Multiple primary breast cancers, first diagnosed between the ages of 50 and 65 y
 An Ashkenazi Jewish individual If criteria 3. An affected or unaffected individual who otherwise does not meet any of the above criteria but with a 2.5%-5% If testing for other probability of *BRCA1/2* pathogenic variant based on prior probability models (eg, Tyrer-Cuzick, BRCAPro, CanRisk)<sup>b</sup> criteria hereditary not met, syndrome There is a low probability (<2.5%) that testing will have findings of documented clinical utility in the following consider not met. scenarios: testing then cancer 1. Women diagnosed with breast cancer at age >65 y, with no close relative<sup>f</sup> with breast, ovarian, pancreatic, or for other screening hereditary as per NCCN 2. Men diagnosed with localized prostate cancer with Gleason Score <7 and no close relative with breast, syndromes ovarian, pancreatic, or prostate cancer Screening Guidelines<sup>†</sup> **Footnotes** on CRIT-2A\*

Taken from Daly et al., 2021.2

CRIT-2


Version Date: 01/30/23

\*Available online, in these guidelines, at NCCN.org. †To view the most recent version of these guidelines, visit NCCN.org

Version 2.2021, 11/20/20 © National Comprehensive Cancer Network, Inc. 2021. All rights reserved.

The NCCN Guidelines® and this illustration may not be reproduced in any form without the express written permission of NCCN.